CLINICAL TRIAL: NCT05357651
Title: A Phase 1, Multicenter, Open-Label Study to Evaluate the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, and Immunogenicity of LB1410, A Recombinant Anti-PD-1 and Anti-TIM-3 Humanized Bispecific Antibody for Injection in Patients With Advanced Solid Tumors or Lymphoma（Keyplus-001）
Brief Title: A Study to Assess the Safety and Efficacy of LB1410 in Participants With Advanced Solid Tumor or Lymphoma（Keyplus-001）
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: L & L Bio Co., Ltd., Ningbo, China (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: LB1410-CHN-Ⅰ-01
Record Dates: First submitted 2022-04-27; First posted 2022-05-03 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Solid Tumor; Lymphoma
MeSH Terms: conditions — Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Dose Escalation (Experimental): Up to 9 dose cohorts will be sequentially enrolled in the dose escalation part using an accelerated titration combined with the standard 3+3 dose escalation algorithm approach.
  Interventions: Drug: LB1410
- Safety Expansion (Experimental): 2-3 doses were initially selected for safety expansion, with patients with advanced solid tumors as the main research population. Each dose cohort is expected to enroll 9-12 patients.
  Interventions: Drug: LB1410
- Exploratory Expansion (Experimental): The Cohort Exploratory Expansion will enroll subjects by cohort at the RP2D dose, and a total of 4 cohorts (cohorts A, B, C, D) are expected.
  Interventions: Drug: LB1410

INTERVENTIONS:
Drug: LB1410 — anti-PD-1 and anti-TIM-3 bispecific antibody

SUMMARY:
This is a Phase I study designed to evaluate if experimental anti-PD-1 and anti-TIM-3 bispecific antibody, LB1410, is safe, tolerable and efficacious in participants with advanced solid tumors or lymphoma.

DETAILED DESCRIPTION:
This first time in patients, open-label, multi-centre study will have LB1410 administered intravenously (IV) to participants with advanced solid tumors or lymphoma. This study will have 2 parts: Part A which will have dose escalation cohorts and Part B which will have the dose expansion cohorts.

ELIGIBILITY:
Inclusion Criteria:

1. Must be ≥ 18 years of age
2. For dose escalation and safety expansion phases only, patient must have histologically or cytologically confirmed advanced and/or metastatic solid tumor malignancies or lymphoma for which standard treatment fails, or no standard treatment is available, or standard treatment is not applicable at this stage
3. Cohort specific inclusion criteria:

   Cohort A: NSCLC patients with histologically confirmed advanced or metastatic NSCLC who have previously failed anti-PD1/anti-PD-L1 antibody and platinum-based chemotherapy, and have not discontinued treatment due to AEs

   Cohort B: NSCLC patients with histologically confirmed advanced or metastatic NSCLC who have failed previous platinum-containing doublet chemotherapy but have not received PD1/PD-L1 antibody therapy；PD-L1 positive

   Cohort C: CRC patients with advanced colorectal cancer who have received no more than 2 lines of systemic therapy in the past; TIM-3≥10%

   Cohort D: Other advanced solid tumors patients who have received no more than two lines of systemic therapy, including but not limited to small cell lung cancer, endometrial cancer, anal cancer, ovarian cancer, head and neck squamous cell carcinoma, gastric adenocarcinoma or gastroesophageal junction cancer patients
4. During the screening period, tumor tissue wax blocks or white slices of pathological biopsy sections shall be provided, or tumor tissue biopsy materials shall be allowed to be collected for PD-L1 and TIM-3 detection
5. Eastern Cooperative Oncology Group Performance Status 0-1
6. Patients with a life expectancy≥12 weeks
7. Must have at least one measurable lesion for assessment by Response Evaluation Criteria in Solid Tumors (RECIST v1.1) or standard criteria for lymphoma (RECIL 2017)
8. Adequate hematological and organ function measured within 7 days prior to first dose
9. Non-pregnant women and willingness of female participants to avoid pregnancy or male participants willing to avoid fathering children through highly effective methods of contraception

Exclusion Criteria:

1. Pregnancy, lactation, or breastfeeding
2. Ongoing or recent (within 5 years) evidence of significant autoimmune disease that required treatment with systemic immunosuppressive treatments
3. Treatment with anti-cancer therapy or investigational therapy within 28 days prior to the first dose of LB1410
4. Patients who have used PD1 monoclonal antibody and TIM3 monoclonal antibody (both simultaneously or sequentially) in the past, and patients who have used one of them alone can be included
5. Immunosuppressive corticosteroid doses (>10 mg prednisone daily or equivalent) within 2 weeks prior to the first dose of LB1410
6. Active infection , including known infection with human immunodeficiency virus (HIV), or active infection with hepatitis B HBV (HBV DNA> 1000 copy/mL or 200 IU/mL) or hepatitis C virus (HCV)
7. Previous malignant disease (other than the target malignancy to be investigated in this trial) within the last 3 years. Subjects with history of cervical carcinoma in situ, superficial, or non-invasive bladder cancer, or basal cell, or squamous cell cancer in situ or other in situ cancers previously treated with curative intent may be included at the judgment of Investigator
8. History of documented allergic reactions or acute hypersensitivity reactions attributed to treatment with antibody therapies in general, or to any of the components of LB1410
9. Symptomatic or uncontrolled brain metastases, spinal cord compression, or leptomeningeal disease requiring concurrent treatment, including but not limited to surgery, radiation, and/or corticosteroids (participants receiving anticonvulsants are eligible)
10. Participant has not recovered (i.e., to <= Grade 1 or Baseline) from radiation- and chemotherapy-induced AEs (except alopecia, peripheral neuropathy, and ototoxicity, which are excluded if ≥ CTCAE grade 3)
11. History of organ transplantation
12. Inadequate recovery from any prior surgical procedure or having undergone any major surgical procedure within 4 weeks prior to the study drug treatment
13. Impaired cardiac function or clinically significant cardiac disease, including any of the following
14. Interstitial lung disease or interstitial pneumonitis, including clinically significant radiation pneumonitis (i.e., affecting activities of daily living or requiring therapeutic intervention)
15. Type 2 diabetes mellitus or type 2 diabetes patients with poor glycemic control.
16. Underlying medical conditions that, in the Investigator's opinion, will make the administration of the study drug hazardous or obscure the interpretation of toxicity determination or adverse events
17. Patients with a history of active tuberculosis infection within 1 year before enrollment
18. Those with a clear history of neurological or mental disorders, such as epilepsy and dementia, and poor compliance
19. Patients with a history of chronic gastrointestinal inflammation, any active inflammation during screening, or grade 3 or above gastrointestinal reaction after previous immunotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-08-12 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2028-12-30 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of treatment-emergent adverse events (TEAEs) | up to 30 days following last dose.
  According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version 5.0.
Incidence and severity of serious adverse events (SAEs) | up to 90 days following last dose.
  According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version 5.0.
AEs of special interest (immune-related AEs) | up to 90 days following last dose.
  Incidence and severity of immune-related AEs.
Incidence of DLTs | in the first 28 days (Cycle 1).
  The DLT for this study is defined according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE), Version 5.0 and will be evaluated in the dose escalation part, the first 28 days (Cycle 1) of treatment.

SECONDARY OUTCOMES:
Serum PK parameters | Up to finished treatment (each cycle is 28 days).
  AUC0-t and so on.
Overall response rate (ORR) | through study completion, an average of 8 months.
  Evaluation Criteria in Solid Tumors (RECIST) v 1.1 and Immunotherapeutics Response Evaluation Criteria in Solid Tumors (iRECIST) and Response Evaluation Criteria in Lymphoma (2017) (RECIL 2017).
Disease control rate (DCR) | through study completion, an average of 8 months.
  Evaluation Criteria in Solid Tumors (RECIST) v 1.1 and Immunotherapeutics Response Evaluation Criteria in Solid Tumors (iRECIST) and Response Evaluation Criteria in Lymphoma (2017) (RECIL 2017).
Progression-free survival (PFS) | through study completion, an average of 8 months.
  Evaluation Criteria in Solid Tumors (RECIST) v 1.1 and Immunotherapeutics Response Evaluation Criteria in Solid Tumors (iRECIST) and Response Evaluation Criteria in Lymphoma (2017) (RECIL 2017).
Duration of response (DOR) | through study completion, an average of 8 months.
  Evaluation Criteria in Solid Tumors (RECIST) v 1.1 and Immunotherapeutics Response Evaluation Criteria in Solid Tumors (iRECIST) and Response Evaluation Criteria in Lymphoma (2017) (RECIL 2017).
Immunogenicity | up to 90 days following last dose.
  Incidence of anti-drug anti-body (ADA) including the number and percentage of participants who develop detectable ADA.

CONTACTS AND LOCATIONS:
Overall Officials: Caicun Zhou, Principal Investigator — Shanghai Pulmonary Hospital, Shanghai, China
Locations (1):
- Shanghai Pulmonary Hospital, Shanghai, Shanghai Municipality, China